CLINICAL TRIAL: NCT06279013
Title: Managing Symptoms and Psychological Distress During Oral Anti-Cancer Treatment
Brief Title: Comparing Telephone Symptom Monitoring Interventions for Managing Symptoms and Psychological Distress During Oral Anti-Cancer Treatment
Acronym: SYMON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NRG-CC012CD; NCI-2023-10831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC012CD (Other: NRG Oncology); NRG-CC012CD (Other: DCP); NRG-CC012CD (Other: CTEP); R01CA279472 (NIH); UG1CA189867 (NIH)
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Counseling; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Cluster randomized
Who Masked: Outcomes Assessor
Masking Description: Interviewers will be blinded to the study arm; IVR is automated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (IVR monitoring) (Active Comparator): Patients receive IVR symptom monitoring calls once a week for 12 weeks, and a summary symptom report is sent to their provider. Call duration is approximately 15 minutes.
  Interventions: Other: Interview; Other: Medical Chart Review; Other: Monitoring; Other: Questionnaire Administration
- Arm II (ATSM, TIPC) (Experimental): Patients receive the Symptom Management and Survivorship handbook and receive IVR symptom monitoring calls for 12 weeks, with summary symptom reports sent to their provider. Call duration is approximately 20 minutes. Patients who report anxious, discouraged, or sad mood items on their monitoring calls for two consecutive weeks between weeks 1 and 4 also receive TIPC calls for up to 8 weeks. TIPC call duration is approximately 30 minutes.
  Interventions: Other: Counseling; Behavioral: Health Education; Other: Interview; Other: Medical Chart Review; Other: Monitoring; Other: Questionnaire Administration

INTERVENTIONS:
Other: Counseling — Receive TIPC
  Other Names: Counseling Intervention
  Arms: Arm II (ATSM, TIPC)
Behavioral: Health Education — Receive handbook
  Arms: Arm II (ATSM, TIPC)
Other: Interview — Ancillary studies
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Monitoring — Receive IVR symptom monitoring
  Other Names: monitor
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
In this clinical trial, symptom monitoring (interactive voice response [IVR] is compared to automated telephone symptom management [ATSM] and telephone interpersonal counseling [TIPC]) for reducing symptom burden and psychological distress (depressive and anxiety symptoms) among people receiving oral anti-cancer treatment. Symptoms are the number one driver of treatment interruptions and unscheduled health services use. To reduce the risk of these events, symptom monitoring and management are necessary. However, these services are not implemented routinely, especially in the community oncology settings. Further, depressive and anxiety symptoms are a key barrier to enacting symptom self-management strategies. IVR is a form of symptom monitoring where patients, when called, enter their symptom ratings over the phone. Their symptom summary is sent to their provider, and patients may be advised to reach out to their oncology provider, based on their symptoms. The ATSM intervention combines IVR assessments with a Symptom Management and Survivorship educational handbook with self-management strategies. Patients receiving ATSM enter their symptom ratings over the phone and have their symptoms reported to their provider, but patients are also directed to the handbook for strategies to manage elevated symptoms. Patients receiving ATSM who report being anxious, discouraged, or sad will also receive TIPC, which targets psychological distress and its connection to social support and interpersonal communication. Information gathered from this study may help researchers learn more about the best ways to manage patient symptoms and improve patient outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test the effectiveness of Automated Telephone System Management (ATSM) + Telephone Interpersonal Counseling (TIPC) versus active control on patient-level outcome of the summary toxicity index of 24 Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) symptoms that include depressive, anxiety, and other symptoms commonly experienced during oral anti-cancer treatment over weeks 1-12 (immediate effect) and 13-17 (sustained effect).

SECONDARY OBJECTIVE:

I. Test the effectiveness of ATSM+TIPC versus active control on patient-level outcome of unscheduled health services over weeks 1-12 and 13-17.

EXPLORATORY OBJECTIVES:

I. Evaluate implementation outcomes at the practice personnel level (physicians, nurses, nurse practitioners, advanced practice providers, physician assistants, medical assistants, pharmacists, social workers, and other behavioral health professionals):

Ia. Feasibility of implementation of the automated telephone symptom monitoring and TIPC at the community oncology practice.

Ib. Perceptions of acceptability of the automated telephone symptom monitoring and TIPC for the community oncology practice.

Ic. Perceptions of appropriateness of the automated telephone symptom monitoring and TIPC for the community oncology practice.

II. Estimate delivery cost of the ATSM+TIPC and active control and cost savings for the ATSM+TIPC versus active control as a result of reduced unscheduled health services use.

III. Estimate the effect of the ATSM+TIPC versus active control on patient-reported financial burden.

IV. Estimate the differences in the effect of the ATSM+TIPC versus active control on the primary and secondary outcomes according to concurrent administration of oral agent with immune checkpoint inhibitor, other targeted infusion therapy, infusion chemotherapy, or radiation therapy.

OUTLINE: Practices are randomized to 1 of 2 arms.

ARM I: Patients receive IVR symptom monitoring calls once a week for 12 weeks, and a summary symptom report is sent to their provider. Call duration is approximately 15 minutes.

ARM II: Patients receive the Symptom Management and Survivorship handbook and receive IVR symptom monitoring calls for 12 weeks, with summary symptom reports sent to their provider. Call duration is approximately 20 minutes. Patients who report anxious, discouraged, or sad mood items on their monitoring calls for two consecutive weeks between weeks 1 and 4 also receive TIPC calls for up to 8 weeks. TIPC call duration is approximately 30 minutes.

After completion of study intervention, patients are followed up during weeks 13-17 and practice personnel are assessed at intake and 12 and 25 months later.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICES: All institutions participating in the practice are National Cancer Institute Community Oncology Research Program (NCORP) affiliates or sub-affiliates.
* PRACTICES: Administer oral therapy to at least 40 patients per year that meet protocol eligibility criteria.
* PRACTICES: Completion and submission of the NRG-CC012CD Letter of Intent (LOI) (posted on the Cancer Trials Support Unit [CTSU] website).
* PRACTICES: Having a social worker licensed in behavioral counseling or other person eligible for behavioral licensing in the practice's state or territory (if licensure is required by state or territory) who can be trained to deliver TIPC or willingness of practice to work with TIPC intervener contracted by the study team. Note: If the practice's social worker or other behavioral health professional is trained to deliver TIPC, they will be compensated for their time training and delivering the TIPC intervention.
* PRACTICE PERSONNEL: Age ≥ 18 years.
* PRACTICE PERSONNEL: Planned to be involved in usual care for at least one enrolled patient during patient's participation in the study.
* PRACTICE PERSONNEL: For a social worker or other behavioral health professional who will deliver TIPC intervention, licensure, or eligibility for licensure in behavioral counseling if required by the state or territory.
* PRACTICE PERSONNEL: The practice personnel must provide study-specific informed consent prior to study entry.
* RETAIN PRACTICE PARTICIPATION: In order to maintain participation in the study, practices must enroll at least 8 patients in the first 6 months (based upon the practice's monthly tracking reports) the practice is open to patient accrual to ensure that the practice can meet the accrual goals. If a practice does not meet this criterion they will be replaced.
* RETAIN PRACTICE PARTICIPATION: Complete monthly forms on actions taken on IVR symptom reports. If fewer than 2 forms are completed in the first 6 months of practice's participation, practice will be replaced.
* RETAIN PRACTICE PARTICIPATION: Participate in monthly study calls for the duration of practice's participation in the study.
* PATIENTS: Starting a new course of an oral anti-cancer agent (the list of agents is posted to the CTSU website) other than sex hormone inhibitors, within 4 weeks after registration or have started an oral anti-cancer agent in the past 8 weeks.
* PATIENTS: All concomitant medications and supportive care treatments are acceptable.
* PATIENTS: Age ≥ 18 years.
* PATIENTS: Able to speak and understand English or Spanish.
* PATIENTS: Access to a telephone and ability to answer questions via telephone in English or Spanish.
* PATIENTS: The patient must provide study-specific informed consent prior to study entry and authorization permitting release of personal health information.

Exclusion Criteria:

* PRACTICES: Active telephone symptom management program at the practice that is beyond symptom and oral agent adherence monitoring.
* PATIENTS: Only receiving treatment with sex hormone inhibitors.
* PATIENTS: Enrollment in the intervention arm of another symptom management trial at intake into the trial. Participation in lifestyle trials with primary outcomes other than symptoms is acceptable.
* PATIENTS: Currently receiving regular behavioral counseling for psychological symptoms. Regular behavioral counseling is defined as at least two counseling sessions with a behavioral health care provider scheduled within the past two months. Patients who completed behavioral counseling within 2 months prior to registration are eligible. Behavioral counseling for issues other than psychological symptoms (e.g., as part of weight loss or smoking cessation program) is not an exclusion criterion.
* PATIENTS: Pregnancy at intake into the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Symptom severity/toxicity index | Up to 12 weeks from the start of therapy (trial interventions)
  Toxicity index across 24 symptoms will be measured using Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events. Linear mixed effects or generalized linear mixed effects models will be used.

SECONDARY OUTCOMES:
Unscheduled health services | Up to 17 weeks from the start of therapy (trial interventions)
  Questions with yes/no responses about each type of unscheduled health service use: hospitalizations, use of urgent care, use of the emergency department. If yes, number of days spent in the hospital, number of times visited urgent care or emergency department are recorded.

OTHER OUTCOMES:
Practice personnel time to address weekly interactive voice response (IVR) symptom reports | Up to 25 months
  Practice personnel time to address weekly IVR symptom reports will be determined based on the checklist of action and standard time to complete each action (e.g., 20 minutes to prescribe a medication). Standard times will be determined based on consensus of practice personnel as discussed during a meeting with practices. Total time will be prorated by the number of patients on trial during each month within each practice.
Automated symptom monitoring and telephone interpersonal counseling (TIPC) delivery at the practice (Feasibility) | Up to 25 months
  Assessed using the 4-item Feasibility of Intervention Measure asked for the automated telephone system and separately for the TIPC. A higher total score indicates greater feasibility.
Practice personnel's actions on symptom reports | Up to 25 months
  Practice personnel will select items for actions taken that includes symptom-related oncology visits, oral agent treatment alterations, prescriptions of supportive care medications, and referrals to supportive care services for each patient.
Treatment fidelity | Up to 25 months
  Treatment fidelity will be assessed using time spent by TIPC interveners in the automated telephone symptom management +TIPC arm and fidelity scores from the checklist that indicates time spent on calls, issues discussed, and any problems encountered for TIPC protocol.
Perceptions of intervention acceptability and appropriateness | Up to 25 months
  Measured using the total score from the Acceptability of Intervention Measure and Intervention Appropriateness Measure, each with 4 questions, with higher scores indicating greater acceptability and appropriateness, respectively.
Cost | Up to 5 years
  Total costs (fixed and variable), including personnel time, fixed costs to develop software, and operating costs for the interventions will be calculated. Cost savings in each arm will be calculated using unadjusted and adjusted rates of hospitalizations and urgent care or emergency department visits based on cost data for the States where participating practices will be located.
Functional Assessment of Chronic Illness Therapy - COmprehensive Score for financial Toxicity (COST) | Up to 17 weeks from the start of therapy (trial interventions)
  The COST is a patient-reported outcome measure that describes the financial distress experienced by cancer patients. It includes 12 items rated on a 5-point Likert type scale. The items are summarized into a total score per scoring instructions.
Concurrent treatment interaction | Up to 17 weeks from the start of therapy (trial interventions)
  Concurrent treatments will be collected. Each concurrent treatment will be analyzed separately for the primary and secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Alla Sikorskii, Principal Investigator — NRG Oncology
Locations (34):
- United States (30):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - CARTI Cancer Center, Little Rock, Arkansas
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Lake Regional Hospital, Osage Beach, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Puerto Rico (4):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan